CLINICAL TRIAL: NCT04180761
Title: Phase II Pilot Study to Reduce the Incidence of Peritoneal Carcinoma After Curative Gastrectomy of Gastric Carcinoma or Adenocarcinoma of Gastroesophageal Transition by Hyperthermic Intraperitoneal Chemoperfusion
Brief Title: Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) in Gastric Cancer
Acronym: ProPeC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No partecipants Enrolled
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProPeC
Record Dates: First submitted 2019-11-07; First posted 2019-11-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2019-11

CONDITIONS: Gastric Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIPEC-Treatment (Experimental): Doxorubicin (15 mg/m²/body surface) Cisplatin (75 mg/m²/body surface) applied as hyperthermic intraperitoneal chemotherapy (HIPEC) at 42.5°C for 60 minutes after the gastrectomy.
  All drugs used are approved.
  Interventions: Drug: intraoperative hyperthermic intraperitoneal chemotherapy (HIPEC)

INTERVENTIONS:
Drug: intraoperative hyperthermic intraperitoneal chemotherapy (HIPEC) — single dose application of hyperthermic intraperitoneal chemotherapy (HIPEC) at 42.5°C for 60 minutes after the gastrectomy

SUMMARY:
This study investigates the effect of a combined therapy with gastrectomy and HIPEC in localized advanced gastric cancer.

DETAILED DESCRIPTION:
An operation and the constant further development of the surgical techniques can not always prevent the recurrence of a tumor of the stomach or the transition from the esophagus to the stomach. As reason for this recurrence, the investigators assume that the tumor was already present at the time of the surgery and has crossed the boundaries of the stomach or free tumor cells are located in the peritoneal cavity, even if they can't be found with the bare eye or imaging methods. Such free tumor cells have the possibility of developing metastases within the abdominal cavity.

An innovative local treatment method is being tested in Tübingen and applied to remove any remaining free tumor cells or very small and invisible residual tumors. These free tumor cells can be determined prior to the start of treatment by peritoneal endoscopy (diagnostic laparoscopy). If these can be identified by lavage of the abdominal cavity there is an increased risk for the development of peritoneal metastases. Therefore, in patients with detected free tumor cells in the lavage water of the abdominal cavity, after the removal of the stomach, should be used once a chemotherapy in the abdominal cavity, which is warmer than the body (intraoperative hyperthermic chemotherapy, HIPEC). In this study the investigators want to demonstrate, that the single administration of intraoperative HIPEC with cisplatin and doxorubicin in addition to routine surgery delays the onset of peritoneal metastases and the additional therapy with its low risks is reasonable.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient
* Positive lavage cytology in staging laparoscopy
* Intraoperative R0- or R1-gastrectomy (Re-evaluation intraoperative)
* Histologically confirmed locally advanced, resectable Adenocarcinomas of the stomach (incl. AEG II-III): >cT3 and/or cN+ and cM0 (none existing solid Peritoneal metastases, Re-evaluation intraoperative)
* Neoadjuvant chemotherapy ≥ 2 cycles

Exclusion Criteria:

* < 18 years
* Existence of contraindications or contraindications against the study medication
* Uncompensated Heart Failure (NYHA III and IV)
* Severe CHD, medically insufficient treatable cardiac arrhythmias, uncontrolled arterial hypertension
* Serum creatinine ≥ 1.5 x the standard value or a Creatinine clearance < 60 ml/min/1.73 m2
* Severe pulmonary dysfunction (COPD, PAH), Pulmonary function test confirmed (IVC < 55 %, DLCO < 40%)
* malignant secondary tumor disease that persists for < 5 years (Exception: in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin)
* Participation in other interventional studies that at the time of the ProPeC study inclusion, still are not finished
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of peritoneal metastases and proportion of patients free from peritoneal metastasis after one year after HIPEC. | one year
  The primary objective of the study is to estimate the effect of a combined therapy with gastrectomy and HIPEC in localized advanced gastric cancer. The primary target is the incidence of peritoneal metastases in CT and the proportion of patients who after one year are free from peritoneal metastasis. The study is intended to provide planning data for a subsequent Phase III study in the form of an RCT.

SECONDARY OUTCOMES:
Overall Survival (OS) | one year
  Overall Survival (OS) measured in years.
Progression-free survival (PFS) | one year
  Progression-free survival (PFS) based on imaging (CT).
Number of participants with treatment-related adverse events as assessed by grading according to CTCAE v5.0 and Clavien-Dindo. | one year
  Expected adverse events (AEs) of particular interest must be recorded from grade ≥ III according to CTCAE v5.0 or postoperative complications according to Clavien-Dindo classification from grade ≥ 3b by AE/ADR reporting.
  Unexpected and expected AEs must be documented and reported as SAE from grade IV according to CTCAE v5.0 or from grade 4-5 according to Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- University Department of General, Visceral and Transplant Surgery, Tübingen, Baden-Wurttemberg, Germany